CLINICAL TRIAL: NCT01214798
Title: Study of the Second Hospital of Qinhuangdao
Brief Title: A Case of Sesamoid Displacement Causing the First Metacarpophalangeal Joint Locking
Acronym: SDL
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: The Second Hospital of Qinhuangdao, The Second Hospital of Qinhuangdao
Other Study IDs: SecondQinhuangdao201010
Record Dates: First submitted 2010-10-02; First posted 2010-10-05 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Primary Disease
Keywords: sesamoid displacement,; metacarpophalangeal joint,; radial condylar ridge of the metacarpal head.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Traumatic sesamoid displacement of the first metacarpophalangeal joint can affect thumb function.

DETAILED DESCRIPTION:
Although occurrence is rare, the mechanism of the displacement is commonly complex and varied. Understanding the mechanism is critical for treatment of the disorder. We herein present a locked thumb MCPJ caused by sesamoid displacement.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic sesamoid displacement

Exclusion Criteria:

* Pathologic sesamoid disorder

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1 person
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chenlin Li, M.D., Study Chair — Second Hospital of Qinhuangdao